CLINICAL TRIAL: NCT00042263
Title: Social and Physical Environments and Health Disparities
Brief Title: Healthy Environments Partnership
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 10936-CP-001
Record Dates: First submitted 2002-07-25; First posted 2002-07-26 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Cardiovascular Health
Keywords: health disparities; social environment; physical environment; racial health disparities

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
The Healthy Environments Partnership was established in October 2000, as a part of the National Institute of Environmental Health Sciences "Health Disparities Initiative." The Healthy Environments Partnership seeks to expand the knowledge base of how social and economic inequalities are linked to disparities in cardiovascular health among residents of Detroit. The Healthy Environments Partnership is a project of the Detroit Community-Academic Urban Research Center. The partners are: Brightmoor Community Center, Butzel Family Center, the Detroit Health Department, Friends of Parkside, Henry Ford Health System, Southwest Counseling and Development Services, Southwest Detroit Environmental Vision and University of Detroit Mercy and the University of Michigan School of Public Health, School of Nursing, and the Institute for Social Research.

ELIGIBILITY:
* Age 25 and older
* Resident of three designated areas of Detroit, MI

Ages: 25 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2002-04

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Public Health, Ann Arbor, Michigan, United States